CLINICAL TRIAL: NCT04635527
Title: A Phase Ib Study to Evaluate the Safety and Efficacy of IBI318 Combined With Conventional TACE (cTACE) as a Perioperative Treatment for Potentially Resected Hepatocellular Carcinoma
Brief Title: A Study on the Safety and Effectiveness of IBI318 Combined With Conventional TACE (cTACE) as a Perioperative Treatment for Potentially Resected Hepatocellular Carcinoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to the company's development strategy adjustment ，Innovent Bioligics decided not to continue the study after consultation with investigators.
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIBI318F101
Record Dates: First submitted 2020-11-13; First posted 2020-11-19 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IBI318 combined with conventional TACE (cTACE) (Experimental)
  Interventions: Drug: IBI318; Procedure: cTACE
- Placebo combined with conventional TACE (cTACE) (Placebo Comparator)
  Interventions: Procedure: cTACE; Drug: placebo

INTERVENTIONS:
Drug: IBI318 — before surgery IBI318 intravenous injection Q2W,after surgery IBI318 intravenous injection Q4W
  Arms: IBI318 combined with conventional TACE (cTACE)
Procedure: cTACE — conventional transarterial chemoembolization
Drug: placebo — before surgery placebo intravenous injection Q2W,after surgery placebo intravenous injection Q4W
  Arms: Placebo combined with conventional TACE (cTACE)

SUMMARY:
The purpose of this phase Ib study is to assess the safety, tolerability and effectiveness of IBI318 in combination with conventional TACE (cTACE) in patients with potentially resected hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years and ≤ 75 years at the time of consent.
2. Hepatocellular carcinoma confirmed by histology/cytology.
3. Lesions with measurable disease at baseline by mRECIST.
4. Barcelona Clinic Liver Cancer stage A or B for hepatocellular carcinoma exceeding Milan criteria.
5. Child-Pugh: <=6
6. Adequate organ and bone marrow function.

Exclusion Criteria:

1. With fibrous lamellar hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, cholangiocarcinoma components in tumor tissues.
2. Having previously received standard systemic therapy, ablative therapy, interventional therapy and surgical treatment for hepatocellular carcinoma.
3. Potential liver transplant candidates
4. Have a history of hepatic encephalopathy or have a history of liver transplantation.
5. With clinical symptoms requires drainage of pleural effusion, ascites or pericardial effusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-12-24 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2023-03-07 (Actual)

PRIMARY OUTCOMES:
Number of participants experiencing clinical and laboratory adverse events (AEs) | Up to 90 days post last dose

SECONDARY OUTCOMES:
The percentage of subjects with pathological Complete Response (pCR) after liver resection | 3 years
The percentage of subjects with major pathological response (MPR) after liver resection | 3 years
The percentage of subjects with R0 resection | 3 years
Objective response rate (ORR) in two arms based on mRECIST by investigator | 3 years
Disease-free survival (DFS) in two arms based on mRECIST by investigator | 3 years
Overall survival (OS) in two arms | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital Zhejiang University, Hangzhou, Zhejiang, China